CLINICAL TRIAL: NCT01833585
Title: Pilot Study of Treatment of Chronic Critical Limb Ischemia With G-CSF-mobilized Autologous Peripheral Blood Mononuclear Cells
Brief Title: Treatment of Chronic Critical Limb Ischemia With G-CSF-mobilized Autologous Peripheral Blood Mononuclear Cells
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIRIRAJR015533013
Record Dates: First submitted 2013-04-09; First posted 2013-04-17 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Critical Limb Ischemia; Atherosclerosis; Ischemic Ulcer; Gangrene
Keywords: critical limb ischemia; atherosclerosis; ischemic ulcer; rest pain; gangrene
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Atherosclerosis; Gangrene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- peripheral blood mononuclear cells (Experimental): peripheral blood mononuclear cells will be injected to calf muscle of critical limb ischemia
  Interventions: Biological: Peripheral blood mononuclear cell

INTERVENTIONS:
Biological: Peripheral blood mononuclear cell — Peripheral blood mononuclear cell solution 59 cc will be injected to the gastrocnemius muscle of ischemic limb of patients with critical limb ischemia

SUMMARY:
The purpose of this study is to determine the safety and efficacy of G-CSF-mobilized autologous peripheral blood mononuclear cell injection to ischemic limbs of patients with critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with critical limb ischemia confirmed by toe pressure, ABI, TCOM
* Levels of arterial occlusion are femoropopliteal or tibioperoneal occlusion
* Poor distal artery runoff
* Age 18-70 year

Exclusion Criteria:

* Planned for major amputation within 4 weeks
* Receive blood component within 4 weeks
* Acute myocardial infarction
* severe valvular heart disease
* renal failure
* liver failure
* Cancer
* Hypercoagulable state
* Severe infection
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of patients without major amputation after mononuclear cell injection | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Nuttawut Sermsathanasawadi, MD.,Ph.D., Principal Investigator — Mahidol University
Locations (1):
- Vascular Surgery, Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand